CLINICAL TRIAL: NCT04980300
Title: Delaware Physical Exercise and Activity for Knee Osteoarthritis (PEAK)
Brief Title: Delaware Physical Exercise and Activity for Knee Osteoarthritis
Acronym: PEAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1730922
Record Dates: First submitted 2021-07-17; First posted 2021-07-28 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: Physical Activity; Physical Therapy; Telehealth; Strengthening Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Virtual consultation sessions with a physical therapist, focusing on lower extremity strengthening exercises, physical activity (i.e., walking), and education about knee osteoarthritis.
  Interventions: Behavioral: Intervention
- Control (Active Comparator): Web-based resources on knee osteoarthritis, including an overview of knee osteoarthritis, brief anatomy of the knee and how that is related to pain, different types of arthritis pain and how to manage it, and how to be active with arthritis.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Participants in the Intervention arm will receive five virtual consultation sessions, delivered by a physical therapist over 12 weeks (at Weeks 1, 2, 4, 7, and 10) and lasting approximately 45-60 minutes each. Each session will focus on lower extremity strengthening exercises, physical activity (i.e., walking), and education about knee osteoarthritis. Participants will be provided with an exercise manual, tracking log, educational manual, and a step counter. Participants will be prescribed up to 6 exercises (quadriceps, hip abductor/gluteal, hamstrings/gluteal, calf, balance) and daily walking step goals. Progression will be a joint decision by the participant and physical therapist. Education will include information on knee osteoarthritis, managing pain, being active, weight loss, dealing with setbacks, and progressing activity. The physical therapist will also discuss barriers and facilitators to meeting and progressing goals as appropriate.
  Arms: Intervention
Behavioral: Control — Participants in the Control arm will receive access to a study-specific website that navigates them to a variety of web-based resources on knee osteoarthritis. Topics for the various resources include an overview of knee osteoarthritis, brief anatomy of the knee and how that is related to pain, different types of arthritis pain and how to manage it, and how to be active with arthritis. Sessions range from 20 - 70+ minutes.
  Arms: Control

SUMMARY:
The objective of this project is to examine the efficacy of an innovative Telehealth Physical Therapy (PT) program for adults with knee osteoarthritis (OA) to increase physical activity over 12 weeks in adults with knee OA compared to a control group receiving web-based resources about knee OA. One hundred individuals with knee osteoarthritis (OA), who are over the age of 45, and are also looking to move more, will be randomized into a brief or expanded intervention group. The control includes an online, guided video orientation from a physical therapist to web resources for strengthening exercises, physical activity, and pain management strategies for knee OA. The intervention includes up to 5 online consultations with a physical therapist over a 12-week period who will prescribe strengthening exercises, physical activity goals, and pain management strategies for knee OA.

DETAILED DESCRIPTION:
Delaware PEAK (Physical therapy Exercise and Activity for Knee osteoarthritis) is a delivered remotely by a physical therapist over 5 one-on-one video conference (Zoom Platform) consultations lasting 45 to 60 minutes each over 12 weeks. Each consultation focuses on strengthening exercises, physical activity goals, and education to debunk common OA-related myths and misconceptions. Delaware PEAK utilizes a well-established behavioral counseling method, Motivational Interviewing, to increase self-efficacy (confidence) related to exercise, while delivering all aspects of the intervention.

The objective of this project is to examine the efficacy of Delaware PEAK to increase physical activity in adults with knee OA compared to a control group receiving web-based resources about knee OA and exercise. The rationale for our study is that there is a need to examine whether PEAK can directly target the mismatch between OA recommendations and practice patterns. Our central hypothesis is that Delaware PEAK will increase physical activity and will increase the belief that exercise is helpful and not harmful, compared with a control group receiving web-based OA treatment resources. Successful completion of this proposal will provide the evidence necessary to scale up this low-cost intervention, with the goal of increasing the number of adults who use exercise to manage their knee OA and thus reducing the burden of disease.

The primary endpoint of our study is to examine the efficacy of a physical therapist-delivered exercise intervention (Delaware PEAK) to increase MVPA over 12 weeks compared to a control group receiving web-based resources about knee OA and exercise.

The secondary analyses endpoint of our study is to examine the efficacy of a physical therapist-delivered exercise intervention (Delaware PEAK) to increase health beliefs in Physical Exercise and Physical Therapy, light physical activity (LPA), and steps per day, over 24 weeks compared to a control group receiving web-based resources about knee OA and exercise. We also will assess change in MVPA over 24 weeks.

Our exploratory endpoints include change in pain, symptoms, function in activities of daily living, function in sport and recreation, and quality of life over 12 weeks and 24 weeks. We will also examine change in treatment expectations before and after randomization. Lastly, we will examine change in treatment adherence from 12 to 24 weeks among those in the expanded intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. meet the National Institute for Health and Care Excellence Osteoarthritis (NICE) clinical criteria:

   1. being at least 45 years of age;
   2. having activity-related joint pain;
   3. having morning stiffness ≤ 30 minutes;
2. have a history of knee pain for at least 12 weeks;
3. are interested in becoming more physically active;
4. have either a cell phone or laptop/desktop computer with broadband internet connection and working email address; and
5. are able to commit to the study for 12 weeks and willing to wear physical activity monitors
6. live in the contiguous United States
7. comfortable participating in a program delivered in English
8. is able to safely participate in a moderate-intensity exercise as determined by a pre-exercise screen questionnaire.

Exclusion Criteria:

1. regularly exercise more than 60 minutes/week; or
2. has a scheduled knee or hip joint replacement; or
3. has had physical therapy for knee OA in the past 6 months; or
4. participated in a strength training program for the lower extremities in the past 6 months.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

REFERENCES:
- [Derived] Aily JB, Copson J, Voinier D, Jakiela J, Hinman R, Grosch M, Noonan C, Armellini M, Schmitt L, White M, White D. Understanding Recruitment Yield From Social Media Advertisements and Associated Costs of a Telehealth Randomized Controlled Trial: Descriptive Study. J Med Internet Res. 2023 May 18;25:e41358. doi: 10.2196/41358. PMID 37200067
- [Derived] Jakiela JT, Voinier D, Hinman RS, Copson J, Schmitt LA, Leonard TR, Aily JB, Bodt BA, White DK. Comparing an Expanded Versus Brief Telehealth Physical Therapist Intervention for Knee Osteoarthritis: Study Protocol for the Delaware PEAK Randomized Controlled Trial. Phys Ther. 2023 Feb 1;103(2):pzac139. doi: 10.1093/ptj/pzac139. PMID 36200390

RESULTS

PARTICIPANT FLOW:
Groups:
- Expanded Intervention: Virtual consultation sessions with a physical therapist, focusing on lower extremity strengthening exercises, physical activity (i.e., walking), and education about knee osteoarthritis.
  Expanded Intervention: Participants in the Expanded Intervention arm will receive five virtual consultation sessions, delivered by a physical therapist over 12 weeks (at Weeks 1, 2, 4, 7, and 10) and lasting approximately 45-60 minutes each. Each session will focus on lower extremity strengthening exercises, physical activity (i.e., walking), and education about knee osteoarthritis. Participants will be provided with an exercise manual, tracking log, educational manual, and a step counter. Participants will be prescribed up to 6 exercises (quadriceps, hip abductor/gluteal, hamstrings/gluteal, calf, balance) and daily walking step goals. Progression will be a joint decision by the participant and physical therapist. Education will include information on knee osteoarthritis, managing pain, being active, weight loss, dealing with setbacks, and progressing activity. The physical therapist will also discuss barriers and facilitators to meeting and progressing goals as appropriate.
- Brief Intervention: Web-based resources on knee osteoarthritis, including an overview of knee osteoarthritis, brief anatomy of the knee and how that is related to pain, different types of arthritis pain and how to manage it, and how to be active with arthritis.
  Brief Intervention: Participants in the Brief Intervention arm will receive access to a study-specific website that navigates them to a variety of web-based resources on knee osteoarthritis. Topics for the various resources include an overview of knee osteoarthritis, brief anatomy of the knee and how that is related to pain, different types of arthritis pain and how to manage it, and how to be active with arthritis. Sessions range from 20 - 70+ minutes.
Period: Baseline to 12 Weeks
Arm/Group | Expanded Intervention | Brief Intervention
Started | 51 | 52
Completed (24-week follow up) | 45 | 51
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 4 | 0
Period: 12 Weeks to 24 Weeks
Arm/Group | Expanded Intervention | Brief Intervention
Started | 45 | 51
Completed | 41 | 46
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Expanded Intervention | Brief Intervention | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.1) | 61.2 (8.0) | 60.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 45 | 85
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 50 | 49 | 99
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  White | 43 | 44 | 87
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kilograms] — Participant weight in kg
  kilograms | 96.4 (23.1) | 95.9 (22.1) | 96.2 (22.5)
Height [Mean (Standard Deviation); unit: Meters] — Study participant height in meters
  Meters | 1.7 (0.1) | 1.6 (0.1) | 1.7 (0.1)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m squared] | 34.4 (7.8) | 35.7 (8.4) | 35.0 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Moderate-to-vigorous Intensity Physical Activity
Description: Actigraph GT3X monitor to be worn over the right hip during waking hours. Participants will be instructed to wear the monitor for 7 consecutive days, and then return the monitor via mail in a pre-addressed, pre-stamped envelope that is provided.
  Units are in minutes/day of Moderate to vigorous intensity physical activity (MVPA), min 0, max 1440, with higher scores representing more time in MVPA
Time Frame: Baseline to 12 weeks as primary outcome Baseline to 24 weeks as secondary outcome
Population: For activity monitor data, we used a modified intention-to-treat method, i.e., all randomly assigned participants who wore the monitor for > 4 days for at least 10 hours/day at baseline were included in analyses. There were 15 (14.6%) study participants who were randomized, but did not have valid baseline activity monitor data despite wearing the monitor and were excluded from the primary analysis. Thus, the modified intention-to-treat sample included n=88.
Measure: Mean (95% Confidence Interval); unit: min/day of MVPA
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 47
min/day of MVPA
  12 weeks - Baseline | 0.7 [-4.8 to 6.2] | 2.6 [-2.6 to 7.7]
  24 weeks - Baseline | 2.7 [-2.9 to 8.2] | 1.6 [-3.6 to 6.8]

2. Secondary Outcome: Change in Treatment Beliefs of Physical Therapy: Positive
Description: Participants will be asked to complete the treatment Beliefs of OA (TOA) Physical Therapy measure, which is a 9-item questionnaire that assesses health beliefs (positive and negative) related to physical therapy.
  Scores of the TOA PT Positive are on a scale of 7 to 28 with higher scores mean better outcome, i.e., more positive treatment beliefs
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat (ITT) sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Brief Intervention
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 1.0 [-0.7 to 2.8] | 0.4 [-2.1 to 1.3]
  24 weeks - Baseline | 0.4 [-1.4 to 2.2] | -0.6 [-2.2 to 1.1]

3. Secondary Outcome: Change in Treatment Beliefs of Physical Exercise: Positive
Description: Participants will be asked to complete the treatment Beliefs of OA (TOA) Physical Exercise measure, which is a 13-item questionnaire that assesses health beliefs (positive and negative) related to physical activity.
  Scores of the TOA PE Positive are on a scale of 7 to 28 with higher scores mean better outcome, i.e., more positive treatment beliefs
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 1.3 [-0.6 to 3.2] | 0.0 [-1.8 to 1.8]
  24 weeks - Baseline | 1.2 [-0.7 to 3.1] | -0.4 [-2.2 to 1.4]

4. Secondary Outcome: Change in Light Intensity Physical Activity (LPA)
Description: Data collected using the ActiGraph GT3x activity monitor will also be used to assess change in minutes/week of LPA between baseline and both follow-up timepoints. Minutes/day of LPA can range from 0 minutes/day to 1,440 minutes/day (24 hours x 60 minutes).
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: min/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 47
min/day
  12 weeks - Baseline | 3.8 [-22.6 to 30.2] | 2.6 [-22.0 to 27.3]
  24 weeks - Baseline | -3.4 [-30.0 to 23.1] | -13.1 [-38.0 to 11.7]

5. Secondary Outcome: Change in Steps/Day
Description: Data collected using the ActiGraph GT3x activity monitor will also be used to assess change in average steps/day between baseline and both follow-up timepoints. Steps/day can be any value greater than or equal to 0. Valid data includes those who wore the ActiGraph for > 4 days.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Steps/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 47
Steps/day
  12 weeks - Baseline | 517.5 [-252.8 to 1287.8] | 259.0 [-462.2 to 980.1]
  24 weeks - Baseline | 269.3 [-505.7 to 1044.4] | -206.5 [-933.6 to 520.5]

6. Secondary Outcome: Change in Treatment Beliefs of Physical Therapy: Negative
Description: Participants will be asked to complete the treatment Beliefs of OA (TOA) Physical Therapy measure, which is a 9-item questionnaire that assesses health beliefs (positive and negative) related to physical therapy.
  Scores of the TOA PT Negative are on a scale of 4 to 16 with higher scores mean worse outcome, i.e., more negative treatment beliefs
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | -0.6 [-1.9 to 0.6] | 1.0 [-0.2 to 2.1]
  24 weeks - Baseline | -1.0 [-2.2 to 0.3] | 0.5 [-0.6 to 1.7]

7. Secondary Outcome: Change in Treatment Beliefs of Physical Exercise: Negative
Description: Participants will be asked to complete the treatment Beliefs of OA (TOA) Physical Exercise measure, which is a 13-item questionnaire that assesses health beliefs (positive and negative) related to physical activity.
  Scores of the TOA PE Negative are on a scale of 4 to 16 with higher scores mean worse outcome, i.e., more negative treatment beliefs
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | -0.6 [-1.9 to 0.6] | 1.0 [-0.2 to 2.1]
  24 weeks - Baseline | -1.0 [-2.2 to 0.3] | 0.5 [-0.6 to 1.7]

8. Other Pre Specified Outcome: Exploratory Outcome: Change in Knee Pain (Visual Analogue Scale)
Description: Change in knee pain will be measured using a single-item Visual Analog Scale (VAS) question in which the participant will indicate their pain in each knee. Scores range from 0-100 where 0 is no pain and 100 is the worst pain imaginable. An index knee to be used for analysis is defined as the knee with worse pain at baseline.
  Scores of the Knee pain Visual Analogue Scale are on a scale of 0 to 100 with higher scores mean worse outcome, i.e., more pain
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | -29.7 [-40.5 to -18.9] | -8.8 [-19.1 to 1.6]
  24 weeks - Baseline | -25.7 [-36.8 to -14.7] | -14.2 [-24.5 to -3.8]

9. Other Pre Specified Outcome: Exploratory Outcome: Change in Knee Injury and OA Outcome Score (KOOS) Pain Subscale
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item questionnaire that assesses five domains, including pain, symptoms (other than pain), function in activities of daily living, function in sport and recreation, and quality of life. The KOOS has subscale scores for Pain, Symptoms, ADL Function, Sport & Recreation Function, and Quality of Life. Scores are transformed to a 0-100 scale with 0 indicating extreme knee problems and 100 indicating no knee problems.
  KOOS Pain, min 0, max 100, with higher scores representing a better outcome
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 10.6 [5.0 to 16.2] | 3.7 [-1.5 to 8.9]
  24 weeks - Baseline | 10.0 [4.3 to 15.6] | 3.8 [-1.5 to 9.0]

10. Other Pre Specified Outcome: Exploratory Outcome: Change in Treatment Expectations
Description: The participant will complete a Treatment Expectations Question, which asks the participant how effective they expect the intervention to be for their knee. This question will be collected at the baseline timepoint: right before and right after randomization. Answers will be expressed as frequencies and percentages for each of the following categories: No effect at all, Minimal improvement, Moderate improvement, Large improvement, and Complete recovery, as well as reported as an increase, decrease, or no change in treatment expectations.
  Score ranges from 1 to 5 with higher scores representing higher expectations of improvement following treatment.
Time Frame: Baseline and after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  Pre-Randomization | 3.1 (0.7) | 3.1 (0.6)
  Post-Randomization | 3.0 (0.7) | 2.6 (0.7)

11. Other Pre Specified Outcome: Exploratory Outcome: Change in Exercise Adherence Rating Scale (EARS)
Description: For the Expanded Intervention, adherence to strengthening exercises and physical activity will be measured using the Exercise Adherence Rating Scale (EARS). The EARS includes 6 items whose total score ranges from 0 to 24, where a higher score indicates greater adherence.
Time Frame: 12 weeks and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: The EARS was only collected in the Intervention Group at 12 weeks and 24 weeks.
  The EARS includes 6 items whose total score ranges from 0 to 24, where a higher score indicates greater adherence and a score of 12 represents neutral agreement to exercise adherence.
Arm/Group | Intervention Group
Number analyzed (Participants) | 45
units on a scale
  12 weeks | 15.1 (6.1)
  24 weeks | 11.1 (6.6)

12. Other Pre Specified Outcome: Exploratory Outcome: Change in Knee Injury and OA Outcome Score (KOOS) Symptoms Subscale
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item questionnaire that assesses five domains, including pain, symptoms (other than pain), function in activities of daily living, function in sport and recreation, and quality of life. The KOOS has subscale scores for Pain, Symptoms, ADL Function, Sport & Recreation Function, and Quality of Life. Scores are transformed to a 0-100 scale with 0 indicating extreme knee problems and 100 indicating no knee problems.
  KOOS Symptoms, min 0, max 100, with higher scores representing a better outcome
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 6.0 [1.2 to 10.9] | 2.2 [-2.4 to 6.8]
  24 weeks - Baseline | 5.8 [0.9 to 10.7] | 0.6 [-4.0 to 5.1]

13. Other Pre Specified Outcome: Exploratory Outcome: Change in Knee Injury and OA Outcome Score (KOOS) ADL Subscale
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item questionnaire that assesses five domains, including pain, symptoms (other than pain), function in activities of daily living, function in sport and recreation, and quality of life. The KOOS has subscale scores for Pain, Symptoms, ADL Function, Sport & Recreation Function, and Quality of Life. Scores are transformed to a 0-100 scale with 0 indicating extreme knee problems and 100 indicating no knee problems.
  KOOS ADL, min 0, max 100, with higher scores representing a better outcome
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 12.5 [6.3 to 18.6] | 4.4 [-1.4 to 10.2]
  24 weeks - Baseline | 9.5 [3.3 to 15.7] | 4.9 [-0.9 to 10.7]

14. Other Pre Specified Outcome: Exploratory Outcome: Change in Knee Injury and OA Outcome Score (KOOS) Sports and Recreation Subscale
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item questionnaire that assesses five domains, including pain, symptoms (other than pain), function in activities of daily living, function in sport and recreation, and quality of life. The KOOS has subscale scores for Pain, Symptoms, ADL Function, Sport & Recreation Function, and Quality of Life. Scores are transformed to a 0-100 scale with 0 indicating extreme knee problems and 100 indicating no knee problems.
  KOOS Sports and Recreation, min 0, max 100, with higher scores representing a better outcome
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 15.2 [2.8 to 27.7] | 4.0 [-7.8 to 15.7]
  24 weeks - Baseline | 7.0 [-5.6 to 19.6] | 3.7 [-8.0 to 15.5]

15. Other Pre Specified Outcome: Exploratory Outcome: Change in Knee Injury and OA Outcome Score (KOOS) Quality of Life Subscale
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42-item questionnaire that assesses five domains, including pain, symptoms (other than pain), function in activities of daily living, function in sport and recreation, and quality of life. The KOOS has subscale scores for Pain, Symptoms, ADL Function, Sport & Recreation Function, and Quality of Life. Scores are transformed to a 0-100 scale with 0 indicating extreme knee problems and 100 indicating no knee problems.
  KOOS Quality of Life, min 0, max 100, with higher scores representing a better outcome
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: We analyzed our intention to treat sample, which included all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 51
units on a scale
  12 weeks - Baseline | 14.4 [7.7 to 21.2] | 5.2 [-1.2 to 11.5]
  24 weeks - Baseline | 15.1 [8.3 to 21.9] | 4.5 [-1.9 to 10.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study enrollment until study completion at the 24 week follow up.
Description: The study team may become aware of an AE through spontaneous report of the patient (e.g., via phone call or email), or through scheduled intervention consultations for participants in the Expanded intervention group. Adverse events were collected from study enrollment until study completion at the 24 week follow up.
Arm/Group | Expanded Intervention | Brief Intervention
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 3/52
Other Adverse Events (participants affected / at risk) | 44/51 | 10/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expanded Intervention (N=51) | Brief Intervention (N=52)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) — Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expanded Intervention (N=51) | Brief Intervention (N=52)
Back (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Hip/Thigh (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Knee (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Ankle/Foot (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Other (Musculoskeletal and connective tissue disorders) | 25 (25) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT04980300/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT04980300/SAP_007.pdf